CLINICAL TRIAL: NCT05973695
Title: Effects of Clamshell Versus Gluteal Bridge Exercises on Low Back Pain, Gluteal Strength and Disability Due to Prolonged Sitting in Females With Gluteal Amnesia
Brief Title: Effects of Clamshell Versus Gluteal Bridge Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0128 UMIA
Record Dates: First submitted 2023-06-27; First posted 2023-08-03 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Lower Crossed Syndrome
Keywords: gluteal weakness; disability; pain; gluteal amnesia
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Clamshell Exercise (Active Comparator): Group A will be treated with baseline treatment and clamshell exercises. Lie on your side with your knees slightly bent and with one leg on top of the other. Keep your feet together and lift your top knee until its parallel with your hip. Lower your knee back to the initial position, repeat, and then switch sides. In 1st week 1 sets 10 repetitions. In 2nd week 2 sets of 10 repetitions. In 3rd and 4th week and onwards 3 sets of 10 repetitions.
  Interventions: Other: clamshell exercise
- Group B: Gluteal Bridge exercise (Active Comparator): Group B will be treated with baseline treatment and Gluteal Bridge exercises. Start flat on your back with your legs bent at a 90-degree angle and feet placed flat on the ground. Make sure your toes are turned outward at 45-degree angles and your knees are facing in the same direction as your toes. Drive down through your feet and push your hips up. You should feel this variation fatiguing the outer portion of your thighs. Make sure you keep your knees over your toes throughout the entire movement. Don't let them move forward over the toes. In a controlled motion, let your hips sink back down toward the ground. This completes 1 repetition. Perform 3 sets of 15 repetitions, or 3 rounds of a 30-second hold.
  Interventions: Other: Gluteal Bridge exercises

INTERVENTIONS:
Other: clamshell exercise — For clamshell exercises, Lie on your side with your knees slightly bent and with one leg on top of the other. Keep your feet together and lift your top knee until its parallel with your hip. Lower your knee back to the initial position, repeat, and then switch sides. In 1st week 1 sets 10 repetitions. In 2nd week 2 sets of 10 repetitions. In 3rd and 4th week and onwards 3 sets of 10 repetitions
  Arms: Group A: Clamshell Exercise
Other: Gluteal Bridge exercises — Start flat on your back with your legs bent at a 90-degree angle and feet placed flat on the ground. Make sure your toes are turned outward at 45-degree angles and your knees are facing in the same direction as your toes. Drive d
  Arms: Group B: Gluteal Bridge exercise

SUMMARY:
Gluteal amnesia is a "condition" where the individual is believed to have lost the ability to contract their gluteal muscles - generally the gluteus maximus, though some report it as the gluteus medius. This can take many different names, such as "dead butt", "sleeping glutes", or glutes that are "turned off".Since the gluteus medius normally helps stabilize the pelvis, gluteal amnesia can lead to lower back pain and hip pain, as well as knee and ankle issues, as the body tries to compensate for the imbalance.

DETAILED DESCRIPTION:
A Randomized controlled trial will be conducted at Jinnah Hospital Physiotherapy Clinic & Boston Physiotherapy and wellness Clinic through consecutive sampling technique on 32 patients which will be allocated through simple random sampling through sealed opaque enveloped into group A & group B. Group A will be treated with clamshell exercises at the frequency of 3 sets with 10 repetitions 3 times/ week with baseline treatment. Group B will be treated with gluteal bridge and baseline treatment. Baseline treatment for both groups will be given Hot pack at low back for 10 minutes and Quadriceps and hamstring stretching 3 times with 30 seconds hold. Outcome measures will be conducted through pain, disability and quality of life questionnaire after 6 weeks. Data will be analyzed during SPSS software version 21. After assessing normality of data by Shapiro -Wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* • Female between the ages of 20 to 40 years

  * Prolonged sitting hours >4 hours.
  * Examination- Symptoms provoked by low back movement.
  * Positive Gluteal strength test
  * Positive SLR for hamstring tightness
  * Positive Thomas test for Rectus femoris tightness.

Exclusion Criteria:

* • Osteoporosis

  * Malignancy
  * Vertebral fractures
  * Pervious or scheduled surgery
  * Trauma
  * Pregnancy
  * Psychological conditions

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2023-10-05 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Numerical Pain Rating scale (NPRS) | upto 4 weeks
  The numerical Pain Rating scale (NPRS) assesses the pain in the gluteal region.
  Pain is assessed using a Numeric pain rating (NPRS). The scale ranges from 0 to 10. 0 indicates "no pain", and 10 indicates "worst Pain.
  mild pain score 1 to 3 moderate pain score 4 to 7 severe pain score with interference with functioning. 8 to 10
Oswestry disability score | upto 4 weeks
  Oswestry Disability score is used to measure low back disability.
  Each ten item is scored from 0 to 5, and the total is added and multiplied by 2. Therefore, the ODI ranges from 0 to 100. A higher score on the ODI indicates a more severe disability caused by LBP.
  Oswestry Disability Index will evaluate disability for disability. This questionnaire will be used to assess disability. It comprises 10 items, 7 related to daily activities, 2 related to pain, and 1 related to concentration. Each item scores from 0 to 5. The total score is expressed as a percentage with higher scores related to more significant disability
Quality of Life EQ-5D | upto 4 weeks
  EQ-5D Health-Related Quality of Life Question checked the quality of life of the patients.
  Descriptive system for health-related quality of life states in adults, consisting of five dimensions (Mobility, Self-care, Usual activities, Pain & discomfort, Anxiety & depression), each with five severity levels described by statements appropriate to that dimension.
  The scale ranges from 100 ('the best imaginable health state' or 'the best health state you can imagine') to 0 ('the worst imaginable health state' or 'the worst health you can imagine'). This is used to obtain a respondent's stated preference values, not to record their own health state.

CONTACTS AND LOCATIONS:
Overall Officials: Samrood Akram, Mphil, Principal Investigator — Riphah International University,Lahore
Locations (1):
- Jinnah hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No